CLINICAL TRIAL: NCT02001584
Title: A Study to Examine the, Safety, Tolerability and Pharmacokinetics Co-Administered Baclofen and Memantine in Obese and Lean, Otherwise Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGH-917-001
Record Dates: First submitted 2013-11-15; First posted 2013-12-05 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers;; Obese, Otherwise Healthy Volunteers
MeSH Terms: conditions — Obesity | interventions — Baclofen; Memantine

ARMS (2):
- Healthy Volunteers (Experimental)
  Interventions: Drug: Baclofen; Drug: Memantine
- Obese, Otherwise Healthy Volunteers (Experimental)
  Interventions: Drug: Baclofen; Drug: Memantine; Drug: Placebo

INTERVENTIONS:
Drug: Baclofen
Drug: Memantine
Drug: Placebo
  Arms: Obese, Otherwise Healthy Volunteers

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics of a predefined dose range of co-administered Baclofen and Memantine in non-obese (Part A) and obese (Part B), otherwise healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged 18 to 45 years inclusive;
2. Subjects with body mass index:

   For Part A: ≥18 kg/m² and ≤25 kg/m²; For Part B: ≥33 kg/m² and ≤40 kg/m².
3. Subjects with a total body weight of ≥50 kg (Part A and Part B);
4. Subjects who are healthy as determined by the Investigator based on pre study medical history, physical examination, vital signs (blood pressure, pulse rate, respiratory rate and body temperature) and 12-lead ECG at screening and each admission;
5. Subjects whose clinical laboratory test results are not clinically relevant and are acceptable to the Investigator at screening and each admission;
6. Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase and bilirubin ≤1.5 x upper limit of normal (ULN);
7. Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening;
8. Subjects who are negative for drugs of abuse and alcohol tests at screening and each admission;
9. Subjects who are non-smokers or who have not smoked or used nicotine-containing products for at least 3 months prior to screening;
10. Subjects with an estimated creatinine clearance ≥100 mL/minute for male subjects or

    ≥90 mL/minute for female subjects (Cockcroft-Gault method) at screening;
11. Subjects who are able and willing to give written informed consent.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Dates: Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of co-administered baclofen and memantine via C-SSRS | From Baseline until Follow-up
Safety and tolerability of co-administered baclofen and memantine via Adverse Events | From Baseline until Follow-up
Safety and tolerability of co-administered baclofen and memantine via Vital Signs | From Baseline until Follow-up
Safety and tolerability of co-administered baclofen and memantine via ECG | From Baseline until Follow-up
Safety and tolerability of co-administered baclofen and memantine via Clinical Laboratory Tests | From Baseline until Follow-up

SECONDARY OUTCOMES:
Pharmacokinetic parameters of co-administered baclofen and memantine via Cmax | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via Tmax | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via AUC | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via MRT | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via CL/F | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via T1/2 | From Baseline until Day 32
Pharmacokinetic parameters of co-administered baclofen and memantine via CLR | From Baseline until Day 32

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, United Kingdom